CLINICAL TRIAL: NCT03736096
Title: Validation of the Molecular Diagnosis of Respiratory Viral Infections on the Sputum of Patients With Cystic Fibrosis
Brief Title: Molecular Diagnosis of Respiratory Viral Infections on Sputum From Cystic Fibrosis Patients
Acronym: MUCOVIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: MUCOVIR (2017-A02380-53)
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cystic Fibrosis; Acute Respiratory Infection
Keywords: cystic fibrosis; sputum; nasopharyngeal swab; viral molecular diagnosis; respiratory infection; expectoration
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sputum and nasopharyngeal swab from expectorant CF participants retained at -80°C
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this project is to evaluate the agreement between nasopharyngeal and sputum specimens in terms of detection of viral infection in Cystic Fibrosis (CF) participants.This is a 12-month national, multicenter prospective study (7 centers). Inclusions concern CF participants (children or adults) with signs of acute respiratory infection seen in consultation or hospitalized in their CF Research Center. A molecular viral multiplex search is performed on both nasopharyngeal and expectoration collected samples for each included participant. Determination of viral detection agreement between the two CF respiratory samples is then performed.

DETAILED DESCRIPTION:
Viral respiratory infections in cystic fibrosis (CF) have a significant impact on the progression of the disease. It is therefore essential to look for these viruses. No recommendations are made for the virological follow-up of CF patients and no optimal strategy for the type of sampling required. In non-CF patients, the search for a viral infection is performed by nasopharyngeal sampling. This method of sampling is invasive and uncomfortable for the patient. In CF patients, sputum, non-invasive sampling, is routinely used for bacterial research and may be used for viral infections to avoid invasive nasopharyngeal sampling in patients whose management is heavy.

After giving consent, both sputum and nasopharyngeal swab are collected for each participant. A record of clinical and biological data is also made at inclusion. A molecular viral search is performed on both samples by a multiplex technique detecting a broad spectrum of respiratory viruses. A bacteriological analysis is carried out on sputum. The molecular results will be interpreted blindly according to the main criterion of evaluation, presence or absence of viral infection.

Comparison of expectoration to nasopharyngeal sampling of CF patients for respiratory virological diagnosis should analyse agreement of the molecular viral detection and position CF sputum as an optimal assay for respiratory viruses with the advantage of not being invasive and in all cases routinely taken for the control and bacterial follow-up.

The promotion of sputum as an ad hoc sampling for viral research and epidemiology would facilitate the establishment of surveillance for viral infections in cystic fibrosis and thereby contribute to the CF register data.

ELIGIBILITY:
Inclusion Criteria:

* participant with Cystic Fibrosis
* participant with sign of acute respiratory infection
* participant able to expectorate

Exclusion Criteria:

* participant not able to expectorate
* participant refusing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: participant living with Cystic Fibrosis disease presenting an acute respiratory infection cared in french pediatric or adult Center
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Concordance of viral type detected in both samples for each participant: sputum and nasopharyngeal swab | Day 1
  Comparison of per participant results of viral molecular detection in both sputum and nasapharyngeal samples: 18 different types of respiratory viruses may be qualitatively detected by Molecular analyses (multiplex PCR) the Outcome Measure results will be reported as number of participants with same virus type in both sample - number participant with different virus detected in the two samples - number of participants with no virus detected in both samples - number of participants with one virus detected in nasapharyngeal and no virus in sputum - number of participant with no virus detected in nasopharyngeal and one virus detected in sputum - and so on for every possible combinations

CONTACTS AND LOCATIONS:
Overall Officials: Sophie VALLET, MD, Principal Investigator — CHU Brest
Locations (11):
- France (11):
  - CHU d'ANGERS, Angers
  - CHU de CAEN, Caen
  - CHU de NANTES, Nantes
  - AP-HP - Hôpital TROUSSEAU, Paris
  - CHRU de Rennes, Rennes
  - Centre de PERHARIDY, Roscoff
  - Hôpital FOCH, Suresnes
  - CHU Toulouse CRCM Pediatrique, Toulouse
  - CHU Toulouse CRCM Adulte, Toulouse
  - CHU Tours, Tours
  - CHU de Tours, Tours